CLINICAL TRIAL: NCT06270212
Title: Complementary Systematic Evaluation of a New Medical Device (STAIRWAY) for Open Airways During Sedation
Brief Title: Medical Device for Airway Patency During Sedation
Acronym: STAIRWAY-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stairway Medical AB (Industry)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CIV-ID 23-08-043797
Record Dates: First submitted 2024-01-24; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2023-10

CONDITIONS: Airway Obstruction; Sedation Complication; Perioperative Complication
Keywords: Airway; Device; Hypoxemia; Propofol; Respiration; Sedation
MeSH Terms: conditions — Airway Obstruction; Hypoxia; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Prospective randomized unpaired, and paired crossover, evaluations of study outcome measures in healthy volunteer study participants (PART A), and prospective randomized unpaired evaluation of study outcome measures in study patients (PART B).
  The number of arms reported below (3) refers to unpaired comparisons (PARTS A-B).
Who Masked: Outcomes Assessor
Masking Description: For practical reasons, study participants, sedationists and study investigators on site cannot be masked to study interventions.
  However, procedural interventionists on site and study investigators scrutinizing study outcome data will be masked to study interventions.
  The number of enrolled study participants reported below (46) refers to evaluable ones.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STAIRWAY (Active Comparator): Unpaired evaluation of STAIRWAY during induction of steady-state sedation in volunteer study participants (PART A), and during induction and maintenance of PS according to SOC in study patients (PART B).
  Interventions: Device: STAIRWAY
- NO DEVICE (Other): Unpaired evaluation of NO DEVICE during induction of steady-state sedation in volunteer study participants (PART A), and during induction and maintenance of PS according to SOC in study patients (PART B).
  Interventions: Device: NO DEVICE

INTERVENTIONS:
Device: STAIRWAY — Evaluation of STAIRWAY (new airway device) during sedation.
  Arms: STAIRWAY
Device: NO DEVICE — Evaluation of NO DEVICE during sedation
  Arms: NO DEVICE

SUMMARY:
OVERALL SYNOPSIS

PART A: Systematic evaluation in spontaneously breathing healthy volunteer study participants

* of cumulative duration of manual measures for airway patency and for mask ventilation with airway device prototype (STAIRWAY) vs. standard procedure (no device) during target-controlled induction of mild and moderate-to-deep sedation with propofol in the supine position
* of minimum anteroposterior and lateral transpharyngeal distances at tongue-base and soft-palate levels, determined by magnetic resonance imaging (MRI) with STAIRWAY vs. biteblock or no device during no, mild and moderate-to-deep steady-state sedation with propofol in the supine position.

PART B: Systematic evaluation (in the body position [normally supine] considered most optimal for the procedural intervention) of the cumulative duration

* of adjuvant manual airway support and ventilation
* of respiratory arrest (interrupted monitoring of endtidal carbon dioxide [ETCO2])
* of hypoxemia (hemoglobin saturation of oxygen [SpO2] <95 %), and
* of perceived sedational comfort, of sedational and procedural usability, and of sedational and procedural preference with STAIRWAY vs. standard procedure (biteblock or no device) during PS according to SOC for scheduled diagnostic or therapeutic procedures planned to be carried out under PS with propofol in spontaneously breathing study patients.

DETAILED DESCRIPTION:
NUMBERS OF STUDY PARTICIPANTS

PART A: 12 (6 female) evaluable study participants (adult healthy volunteers).

PART B: 34 evaluable study participants (adult patients).

DURATION OF INVESTIGATION FOR COLLECTION OF STUDY DATA

PART A: Two months (February until March 2024).

PART B: Six months (February until July 2024).

STUDY FOLLOW-UP

PART A: Short-term questionnaire-based follow-up by individual study participants' survey at study site immediately after appropriate awakening from, and completed collection of study data during, mild and moderate-to-deep steady-state sedation.

PART B: Short-term questionnaire-based follow-up by individual study patients', sedationists' and procedural interventionists' surveys at the study site immediately after appropriate awakening from, and completed collection of study data during, PS according to SOC.

PRIMARY STUDY OBJECTIVES

PART A: Randomized paired crossover comparison of MRI-derived minimum anteroposterior and lateral transpharyngeal distances at tongue-base and soft-palate levels during spontaneous breathing of pure oxygen at mild (Observer Assessment of Alertness/Sedation [OAA/S] level 4) and moderate-to-deep (OAA/S level 2-3) sedation - assessed by estimated target organ levels of propofol according to computerized infusion pump settings, and by bedside judgements of OAA/S levels - in the supine body position with STAIRWAY vs. standard procedure (biteblock or no device).

PART B: Randomized unpaired comparison (by continuous systematic observation and recording) of cumulative duration of adjuvant use of manual airway support and ventilation with STAIRWAY vs. standard procedure (no device) during PS according to SOC - assessed by estimated target tissue levels of propofol according to computerized infusion pump settings, by clinical bedside judgements of sedation levels according to OAA/S, and by monitored Bispectral Index Score (BIS) levels - for scheduled diagnostic or therapeutic procedures planned to be carried out under PS with propofol in the body position (normally supine) most optimal for the procedure.

SECONDARY STUDY OBJECTIVES

PART A: Randomized unpaired comparison of cumulative duration of interrupted ETCO2 monitoring, of SpO2 <95 %, and of adjuvant manual airway measures and mask ventilation, with STAIRWAY vs. no device during computerized target-controlled intravenous (iv) infusion (TCI) of propofol to attain mild and moderate-to-deep steady-state levels of sedation. Individual questionnaire-based evaluation of perceived sedational comfort (VAS units).

PART B: Randomized unpaired comparison of incidence and cumulative duration of interrupted ETCO2 monitoring, and of SpO2 <95 %, during PS according to SOC - assessed by algorithm-based estimated target organ levels of propofol, and by clinical bedside judgements of sedation levels according to OAA/S - for scheduled diagnostic or therapeutic procedures planned to be carried out under PS with propofol in the body position (normally supine) most optimal for the procedure with STAIRWAY vs. no device (standard procedure). Individual questionnaire-based evaluation of perceived sedational comfort (VAS units) by unblinded study patients, of perceived sedational usability (VAS units) by unblinded sedationists, and of perceived procedural conditions (VAS units) by blinded interventionists, soon after completion of PS according to SOC with STAIRWAY or no device.

ELIGIBILITY:
INCLUSION CRITERIA:

PART A: Adult (18-65 years). No known allergy or hypersensitivity to drugs used for routine sedation or to materials (PP or EVA) comprising STAIRWAY. Medically healthy with no comorbidity according to careful investigation by senior anaesthesiologist in charge of the sedation. No in situ magnetic device or implant. No cognitive or psychosocial distress, particularly including claustrofobia. Complete dentation. No mobile teeth, mobile reconstructions or orthodontic braces. Non-pregnant. No ongoing breast-feeding. Ability to communicate in Swedish. Oral and written informed consent to inclusion as healthy volunteer study participant.

PART B: Adult (18 years and above) scheduled for elective diagnostic or therapeutic procedures under PS with propofol. No known allergy or hypersensitivity to drugs used for PS or to materials (PP or EVA) comprising STAIRWAY. Medical comorbidity corresponding to ASA class I-III. No cognitive or psychosocial distress. Complete or partial dentation. No mobile teeth, mobile reconstructions or orthodontic braces. Ability to communicate in Swedish. Oral and written informed consent to inclusion as study participant.

EXCLUSION CRITERIA:

PARTS A-B: Withdrawal of informed consent. Suspected or manifest unforeseen severe allergic reaction. Inability to obtain enough useful study data for practical or medicotechnical reasons.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Transpharyngeal distance during moderate-to-deep steady-state sedation. | Five months
  Differences in minimum anteroposterior and lateral transpharyngeal distances (mm) at tongue-base and soft-palate levels, determined by an experienced radiologist with specific MRI competence, based on MRI scans obtained with a General Electric SIGNA™ Architect 3T MRI scanner, between use of STAIRWAY vs. NO DEVICE during moderate-to-deep (OAA/S level 2-3) steady-state sedation with propofol [PART A].
Duration of manual airway support during PS for clinical procedures. | Six months
  Difference in cumulative duration (s) of adjuvant manual measures for airway support between use of STAIRWAY vs. NO DEVICE during procedural sedation with propofol according to standard of care for scheduled diagnostic or therapeutic procedures planned to be carried out under procedural sedation with propofol [PART B].

SECONDARY OUTCOMES:
Transpharyngeal distance during mild steady-state sedation. | Five months
  Differences in minimum anteroposterior and lateral transpharyngeal distances (mm) at tongue-base and soft-palate levels, determined by an experienced radiologist with specific MRI competence, based on MRI scans obtained with a General Electric SIGNA™ Architect 3T MRI scanner, at tongue-base and soft-palate levels, between use of STAIRWAY vs. NO DEVICE during mild (OAA/S level 4) steady-state sedation with propofol [PART A].
Duration of interrupted capnometric monitoring during sedation. | Six months
  Differences in cumulative duration (s) of interrupted ETCO2 monitoring between STAIRWAY vs. NO DEVICE during induction of mild and moderate-to-deep levels of sedation (Philips Expression MR400 monitor) with propofol [PART A], and during induction and maintenance of procedural sedation with propofol according to standard of care (Philips MX800 monitor) for scheduled diagnostic or therapeutic procedures planned to be carried out under procedural sedation with propofol [PART B].
Duration of manual airway support during induction of steady-state sedation. | Five months
  Differences in cumulative duration (s) of manual measures for adjuvant airway support between STAIRWAY vs. NO DEVICE during induction of mild and moderate-to-deep steady-state sedation with propofol [PART A].
Sedational comfort | Six months
  Perceived sedational comfort, individually assessed by study participants between 0.0 (minimum score) and 10.0 (maximum score) on a 100 mm visual analogue score line, with STAIRWAY or NO DEVICE, after induction of mild and moderate-to-deep steady-state sedation with propofol [PART A], and after procedural sedation with propofol according to standard of care for scheduled diagnostic or therapeutic procedures planned to be carried out under procedural sedation with propofol [PART B].
Conditions for sedation | Six months
  Perceived conditions for sedation, individually assessed by sedationists between 0.0 (minimum score) and 10.0 (maximum score) on a 100 mm visual analogue score line, and individual preference, with STAIRWAY or NO DEVICE, after procedural sedation with propofol according to standard of care for scheduled diagnostic or therapeutic procedures planned to be carried out under procedural sedation with propofol [PART B].
Conditions for procedural intervention | Six months
  Perceived conditions for procedural intervention, individually assessed by interventionists/surgeons between 0.0 (minimum score) and 10.0 (maximum score) on a 100 mm visual analogue score line, and individual preference, with STAIRWAY or NO DEVICE, after procedural sedation with propofol according to standard of care for scheduled diagnostic or therapeutic procedures planned to be carried out under procedural sedation with propofol [PART B].

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Åkeson, Professor, Principal Investigator — Lund University, Malmö, Sweden
Locations (1):
- Skåne University Hospital, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No